CLINICAL TRIAL: NCT02113943
Title: Etude Comparative Monocentrique, randomisée, en Cross-over, en Double Aveugle, Contre Placebo, de l'Action du Citalopram Sur Les paramètres Cognitifs de la Motivation
Brief Title: Double Blind Randomized, Monocentric, Cross-over, Placebo-controlled Study to Evaluate the Effect of Citalopram on Motivation
Acronym: MBBCitalopram
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Model: Crossover | Masking: Triple
Other Study IDs: C13-03; 2013-003496-35 (EudraCT Number)
Record Dates: First submitted 2014-04-07; First posted 2014-04-15 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: Normal Volunteers
MeSH Terms: interventions — Citalopram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Citalopram 30mg

SUMMARY:
The aim of the current study is to examine the role of serotonin on the cognitive parameters of motivation. They are embedded in a conceptual framework of motivation that merges decision-making and reinforcement learning theories. Every action is conceived as path from one state to another. The different states are associated to different values (positive for rewards and negative for punishments), and the different actions to different costs (risk, effort and delay). The tasks are designed such that the sensitivity to the state and action parameters can be inferred by fitting computational models.The primary objective is to characterize the effect of Citalopram 30mg on reward sensitivity, assessed in an incentive force task, in which participants are asked to squeeze a hand grip to win monetary rewards. Secondary objectives are to characterize the effect of Citalopram 30mg on other cognitive parameters of motivation (assessed with a motivational battery that includes rating, choice and learning tasks).

ELIGIBILITY:
Inclusion Criteria:

* Man or woman, age ≥ 18 and < 50
* Weight between 50 kg and 90 kg.
* No contraindication to effort
* No evolutive pathology that could interfere with the current study signed consent
* medical insurance ("sécurité sociale")

Exclusion Criteria:

* Age < 18 or > 50
* Smokers
* Person under curatorship, or guardianship, or with civil rights deprivation
* History of neurologic or psychiatric pathology
* Presence of any psychotropic treatment
* Chronic or actual consumption of alcohol, or psychotropic drugs
* pregnancy, breastfeeding
* Woman of childbearing potential without effective contraception
* Hypersensitivity to atomoxetine or other constituents of the product
* Pheochromocytoma
* Narrow angle Glaucoma
* Liver failure
* Severe Cardiovascular Disorders
* Severe Cerebrovascular Discorders
* Treatment with non-selective Monoamine Oxidase Inhibitor (MAOI) : iproniazide.
* Treatment with Linezoline, Lithium, Milleperthuis, Tramadol, tryptans.
* Treatment with Pimozide, or treatment that can induce a QT prolongation (neuroleptics, class IA and III antiarrythmic, moxifloxacine, erythromicine, methadone, mefloquine, tricyclic antidepressants, lithium, cisapride), or treatment that can induce an hydroelectrolytic inbalance (thiazide diuretics).
* Treatment with Anticoagulants
* Treatment that can decrease seizure threshold: antidepressants, neuroleptics, mefloquine, buproprione, tramadol
* Enzyme inducers, (rifampicine, …)
* Treatment that can interfere with the performance of the subject: beta2 adrenergic agonists, analgesics, corticosteroïds, anti-inflammatory drugs, …

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2014-04; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Reward sensitivity | Multiple Time Frame: 2h after placebo, 2h after Citalopram 30mg
  Apathy will be assessed as the sensitivity to rewards in an incentive force task.
  The primary Outcome measure is the change in this parameter between the placebo condition and the Citalopram condition.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Christophe Corvol, MCU-PH, Principal Investigator — CIC Neurologie GH Pitié Salpêtrière
Locations (1):
- CIC Neurologie GHPS, Paris, France